CLINICAL TRIAL: NCT03662620
Title: A Randomized, Open-label, Single Dose, Replicate Crossover Clinical Trial to Compare the Safety and Pharmacokinetics of YH22162 in Healthy Volunteers
Brief Title: Clinical Trial to Compare the Safety and Pharmacokinetics of YH22162 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YH22162-103
Record Dates: First submitted 2018-09-03; First posted 2018-09-07 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Amlodipine; Chlorthalidone; Drug Evaluation

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, single-dose, 2-treatment, 2-sequence, 4-period replicate crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM1 (Experimental): In ARM1, 32 subjects will be assigned and the subjects will be administered "comparator drug" at Day1/Day43 and "study drug" at Day22/64.
  Interventions: Drug: Telmisartan 80mg + Amlodipine 5mg + Chlorthalidone 25mg
- ARM2 (Experimental): In ARM2, 32 subjects will be assigned and the subjects will be administered "study drug" at Day1/Day43 and "comparator drug" at Day22/64.
  Interventions: Drug: Telmisartan 80mg + Amlodipine 5mg + Chlorthalidone 25mg

INTERVENTIONS:
Drug: Telmisartan 80mg + Amlodipine 5mg + Chlorthalidone 25mg — White colored oval three-layer tablet
  Other Names: Study drug
Drug: Telmisartan 80mg + Amlodipine 5mg + Chlorthalidone 25mg — White and pink colored oval two-layer tablet
  Other Names: Comparator drug

SUMMARY:
This is a phase 1, randomized, open label, single-dose, replicate crossover clinical trial to compare the safety and pharmacokinetics of YH22162 in healthy male volunteers.

Hypothesis: Study drug and comparator drug are showing equal pharmacokinetics.

DETAILED DESCRIPTION:
In ARM1, 32 subjects will be assigned and the subjects will be administered "comparator drug" at Day1/Day43 and "study drug" at Day22/64.

In ARM2, 32 subjects will be assigned and the subjects will be administered "study drug" at Day1/Day43 and "comparator drug" at Day22/64.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male with body mass index(BMI) between 18.5 and 30 kg/m2
* Who has not suffered from clinically significant disease
* Provision of signed written informed consent

Exclusion Criteria:

* History of and clinically significant disease
* Administration of other investigational products within 3 months prior to the first dosing
* Volunteers considered not eligible for the clinical trial by the investigator due to reasons including laboratory test results, ECGs, or vital signs

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2018-12-08 (Actual); Study Completion 2018-12-22 (Actual)

PRIMARY OUTCOMES:
AUClast of Telmisartan/amlodipine/chlorthalidone | 0-168 hrs
  AUClast
Cmax of Telmisartan/amlodipine/chlorthalidone | 0-168 hrs
  Cmax

SECONDARY OUTCOMES:
AUCinf of Telmisartan/amlodipine/chlorthalidone | 0-168 hrs
  AUCinf
Tmax of Telmisartan/amlodipine/chlorthalidone | 0-168 hrs
  Tmax
t1/2 of Telmisartan/amlodipine/chlorthalidone | 0-168 hrs
  t1/2

CONTACTS AND LOCATIONS:
Overall Officials: Mingul Kim, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollanam-do, South Korea

IPD SHARING:
Plan to Share IPD: No